CLINICAL TRIAL: NCT01631370
Title: The Effects of Renal Sympathetic Denervation on Insulin Sensitivity in Patients With Resistant Essential Hypertension
Brief Title: The Effects of Renal Denervation on Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Ulla Kampmann Opstrup, MD, PhD, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKOM20110071
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2015-04

CONDITIONS: Treatment Resistant Essential Hypertension; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal denervation (Experimental): The patients will be examined prior to renal denervation and 6 months after. Thus the patients are their own controls.
  Interventions: Procedure: Renal denervation

INTERVENTIONS:
Procedure: Renal denervation — The patients are examined prior to and 6 months after renal denervation. On the day of examination the patients will have blood samples taken and the hyperinsulinemic euglycemic clamp and muscle and adipose tissue biopsies will be performed.

SUMMARY:
Renal sympathetic nerves contribute to development of hypertension. Sympathetic overactivity also induces insulin resistance and it could therefore be assumed that a renal denervation might improve insulin sensitivity. Studies have shown that glucose metabolism is improved in patients with treatment resistant essential hypertension both 1 and 3 months after renal denervation compared to a control group with treatment resistant essential hypertension. Fasting glucose, insulin and C-peptide decreased significantly as did insulin resistance assessed by HOMA-IR. The investigators wish to investigate the effect of renal denervation on insulin sensitivity using the gold standard - the hyperinsulinemic euglycemic clamp and to investigate the degree of insulin resistance in muscle, liver and adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Systolic daytime ambulatory BP at least 145 mmHg and compliance to a minimum of 3 antihypertensive drugs, including a diuretic

Exclusion Criteria:

* Diabetes
* Pregnancy
* Non compliance
* Heart Failure (NYHA 3-4)
* LV ejection fraction < 50 %
* Renal insufficiency (eGFR<30)
* Unstable coronary heart disease
* Coronary intervention within 6 months
* Myocardial infarction within 6 months
* Claudication
* Orthostatic syncope within 6 months
* Secondary Hypertension
* Permanent atrial fibrillation
* Significant Heart Valve Disease
* Clinically Significant abnormal electrolytes, haemoglobin, Liver enzymes, TSH
* Second and third degree heart block
* Macroscopic haematuria
* Proximal significant coronary stenosis
* Renal artery anatomy not suitable for renal artery ablation (Stenosis, small diameter < 4 mm, length < 2 cm, multiple renal arteries, severe calcifications)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03-30 (Actual); Study Completion 2016-03-03 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity expressed as an M-value | 4 hours
  To assess insulin sensitivity the hyperinsulinemic euglycemic clamp is used. The patients are given 0.8 mU/kg/min insulin as an infusion for 2 hours and the blood glucose is clamped at 5 mmol/l. For assessment of endogenous glucose production (EGP) during the glucose clamps, a tracer (3-3 H glucose) is added to the glucose infusion. The patients will be examined by the hyperinsulinemic euglycemic clamp prior to the renal denervation and 6 months after.

SECONDARY OUTCOMES:
Insulin signaling | 6 months
  Two biopsies from the lateral vastus muscle and two biopsies from the abdominal subcutaneous adipose tissue are obtained under local anesthesia. Biopsies are taken at baseline and during the clamp. Protein expression involved in the insulin signalling cascade is assessed using standard western blotting techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Per Løgstrup, MD Dr Sci, Principal Investigator — Department of Endocrinology and Internal Medicine, Aarhus University Hospital
Locations (1):
- Medical Research Laboratories, Aarhus University Hospital, Aarhus, Denmark